CLINICAL TRIAL: NCT04275466
Title: A Randomized Controlled Trials on the Effect of Necrotic Cavity Lavage After Laparoscope-assisted Debridement for Patients With Infected Pancreatic Necrosis
Brief Title: Perform Necrotic Cavity Lavage or Not After Debridement of Infected Pancreatic Necrosis
Acronym: NCLAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lifei
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-02

CONDITIONS: Pancreatitis,Acute Necrotizing; Pancreas Necrosis
Keywords: acute pancreatitis; infected pancreatic necrosis; laparoscope-assisted debridement; necrotic cavity lavage
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- necrotic cavity lavage (Experimental): This arm was performed necrotic cavity lavage after debridement
  Interventions: Procedure: necrotic cavity lavage
- non-necrotic cavity lavage (No Intervention): This arm was not performed necrotic cavity lavage after debridement

INTERVENTIONS:
Procedure: necrotic cavity lavage — 1. At least two 30- to 36-Fr drainage tubes will be placed into each necrotic cavity. One of these drainage tubes will be used as the lavage tube; the other tube is designed for drainage.
  2. Lavage will begin on the first day after debridement, and the relevant indices will be evaluated every 7 days to decide whether to continue the lavage.
  3. 1200 mL of normal saline will be lavaged into each necrotic cavity every day at a speed of 200 mL/h for 3 hours each time and for a total of two times. The start times of lavage will be 08:00 and 20:00.
  4. The lavage and drainage volumes of the first hour and second hour of each lavage session will be calculated. The lavage of the next hour will be stopped if the lavage volume minus the drainage volume is >100 mL.
  5. Lavage will be suspended if abdominal pain and distention occur, the maximum body temperature is >38.5ºC, or the abdominal pressure is ≥15 mmHg during the lavage procedure.
  Arms: necrotic cavity lavage

SUMMARY:
The infected pancreatic necrosis (IPN) should be treated by debridement and drainage. In recent years, the results of clinical research show that minimally invasive debridement such as video-assisted (laparoscope, nephroscope, endoscopy, etc.) and total laparoscopic debridement can significantly improve the prognosis of IPN patients. After a long period of clinical practice, laparoscope-assisted debridement was selected as the main surgical method in our center. In many large-scale clinical studies, patients after surgery underwent necrotic cavity lavage (such as small omental sac lavage, retroperitoneal space lavage, peripancreatic lavage, etc.), but its necessity and clinical significance were not clearly stated in the guidelines. At present, the clinical research mainly focuses on the improvement of minimally invasive debridement, and less on the necessity of lavage. In the past, necrotic cavity lavage was performed in IPN patients, but long-term clinical observation showed that lavage may lead to spread of infection and increase the incidence of lower extremity venous thrombosis which is not accorded with ERAS(Enhanced Recovery After Surgery). Therefore, since 2012, our center has stopped necrotic cavity lavage for IPN patients after debridement. We retrospectively analyzed the therapeutic effect from February 2014 to August 2017 and found that even without necrotic cavity lavage, better therapeutic effect could be achieved. Meanwhile it can simplify the operation process and avoid infection spread. This treatment method provides a new idea. However, it is a retrospective study not a randomized controlled trials(RCT) which is low effectiveness of proof. Therefore, we design this RCT to verify the necessity of necrotic cavity lavage after laparoscope-assisted debridement for patients with infected pancreatic necrosis.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of IPN
2. onset time of >4 weeks
3. performance of LAD for IPN
4. provision of written informed consent

Exclusion Criteria:

1. the highest temperature in 24 hours of ≥38.5ºC
2. new organ failure occurring within 24 hours after the operation
3. digestive tract fistula, biliary tract or digestive tract obstruction, or bleeding occurring within 24 hours after the operation
4. abdominal pressure of ≥10 mmHg within 24 hours after the operation
5. traumatic pancreatitis or a pancreatic fistula-related infection after the pancreatic operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-06-12 (Estimated); Study Completion 2021-10-12 (Estimated)

PRIMARY OUTCOMES:
sum rate of mortality and major complications | 1 year
  number of deaths and major complications (new organ failure or intraperitoneal hemorrhage/gastrointestinal fistula requiring surgical treatment)/total enrollment

SECONDARY OUTCOMES:
physiological parameter | through study completion, an average of 2 months
  body temperature in degree centigrade
physiological parameter | through study completion, an average of 2 months
  abdominal pressure in mmHg
assay index | through study completion, an average of 2 months
  white blood cell in 109/L
assay index | through study completion, an average of 2 months
  c-reactive protein in mg/L
assay index | through study completion, an average of 2 months
  procalcitonin in ng/ml
assay index | through study completion, an average of 2 months
  interleukin-6 in pg/ml
incidence of peritonitis and lower extremity deep vein thrombosis | through study completion, an average of 2 months
  postoperative complication
Acute Physiology and Chronic Health Evaluation (range:0-71) | through study completion, an average of 2 months
  The score shows the severity of the patients and higher scores mean a worse outcome
Total stay in hospital | through study completion, an average of 2 months
  The time for the patient staying in hospital measured in days
Length of stay in Intensive Care Unit | through study completion, an average of 2 months
  The time for the patient staying in Intensive Care Unit measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No